CLINICAL TRIAL: NCT06072885
Title: Prospective Observational Evaluation of Perioperative Lung Ultrasound Scores in Laparoscopic Pediatric Surgeries
Brief Title: Evaluation of Perioperative Lung Ultrasound Scores in Laparoscopic Pediatric Surgeries
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meltem Savran Karadeniz, MD, Assoc Prof, Istanbul University
Other Study IDs: 2023/796
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Postoperative Pulmonary Atelectasis
Keywords: pediatric anesthesia; Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Laparoscopic pediatric surgery: Pediatric patients who are scheduled for laparoscopic surgeries in supine position (e.g. laparoscopic appendectomy, laparoscopic cholecystectomy, laparoscopic nissen fundoplication)
  Interventions: Other: Lung Ultrasound Scoring

INTERVENTIONS:
Other: Lung Ultrasound Scoring — Pediatric Laparoscopic Surgery patients will be undergone Lung Ultrasound Scoring (LUS) at multiple times perioperatively. LUS is a pragmatic calculation reflecting lung aeration. Thorax is divided into 12 areas, and in every one of them LUS is applied to observe the lung condition. For that, if there are B-lines less than 4 in one area, it is scored as 1 point. For the areas containing more than 3 B-lines, it is scored as 2 points, and if there is any distortion on the pleural line, it is scored as 3 points. The areas with no B-lines is scored as 0 points. Considering these details, lungs with best conditions will reflect 0 points whereas the worst condition lungs will reflect 36 points. LUS will be performed after intubation, before extubation, and after 30th minute in the post anesthesia care unit

SUMMARY:
Laparoscopic surgeries require carbon-dioxide into the abdomen which may occasionally lead to atelectasis. The extent of this atelectasis is not well documented in peri-operative period although it has been extensively researched in critical care set up. In this study, it is aimed to observe the ultrasonographic condition of lungs in laparoscopic pediatric surgeries. The hypothesis was the Lung Ultrasound Scores would worsen in those surgeries by the end of the operation. Aged between 1-18 years pediatric patients who are scheduled for laparoscopic surgeries will be included in the study to observe the changes in the lung visuals throughout the operation. For that, after safe endotracheal intubation first ultrasonography will be performed for the first (T1) time, and the second ultrasonography will be performed once the surgery is finished and before extubation (T2). Lastly, the third evaluation will be performed after 30 minutes in post anesthesia care unit (T3). Lung Ultrasound Score (LUS) is calculated as follows: Both hemi-thoraxes are divided into 6 different zones, and depending on the number of B-lines, which happens due to aeration loss in lung tissue, every zone is scored. If there is no B-line, it is zero points. If the B-lines in the visual lower than 4, the area is scored as 1 point. The areas with B-lines more than 3 is scored as 2 points. Furthermore, if there is any disruption on the pleural face, then the area is scored as 3 points. Accordingly, the worst case scenario refers 36 points, meaning the less the points the better the lung aeration.

Primary outcome is defined as T2 LUS which will show the actual condition of at the end of the surgery. For that, T1 scores and T2 scores will be compared. The secondary outcomes include T3 LUS, (T3-T1)LUS, intraoperative hemodynamics, length of stay in Post Anesthesia Care Unite, postoperative aldrete scores for discharging to ward, and intraoperative ventilation variables.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic pediatric surgeries
* Aged between 1-18 years

Exclusion Criteria:

* Patients with Constitutional lung diseases
* Patients with Heart failure
* Patients with pulmonary hypertension

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients who are scheduled for laparoscopic abdomen surgeries that will be performed in supine position
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Lung Ultrasound Score in T2 time point (After surgery finish, before extubation) | Up to 4 hours
  LUS is a pragmatic calculation reflecting lung aeration. Thorax is divided into 12 areas, and in every one of them LUS is applied to observe the lung condition. For that, if there are B-lines less than 4 in one area, it is scored as 1 point. For the areas containing more than 3 B-lines, it is scored as 2 points, and if there is any distortion on the pleural line, it is scored as 3 points. The areas with no B-lines is scored as 0 points. Considering these details, lungs with best conditions will reflect 0 points whereas the worst condition lungs will reflect 36 points. T2 LUS will be compared to T1 LUS to observe possible significant change in lung condition.

SECONDARY OUTCOMES:
Lung Ultrasound Score in T3 time point (30 minutes after admission to post anesthesia care unit | Up to 4 hours
  To measure Thorax is divided into 12 areas, and in every one of them LUS is applied to observe the lung condition. For that, if there are B-lines less than 4 in one area, it is scored as 1 point. For the areas containing more than 3 B-lines, it is scored as 2 points, and if there is any distortion on the pleural line, it is scored as 3 points. The areas with no B-lines is scored as 0 points. Considering these details, lungs with best conditions will reflect 0 points whereas the worst condition lungs will reflect 36 points. T3 LUS will be compared to T1 LUS to observe possible significant change in lung condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No